CLINICAL TRIAL: NCT04440956
Title: Positron Emission Tomography (PET) Imaging of Patients With Low & Intermediate Grade Neuroendocrine Tumors Using 64Cu-SARTATE: A Single Centre, Open-Label, Non-Randomized, Phase-0 Microdosing Investigation
Brief Title: An Imaging Study of 64Cu-SARTATE Using Positron Emission Tomography in Patients With Neuroendocrine Tumours
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Clarity Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CL01
Record Dates: First submitted 2020-06-11; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — 64Cu-SARTATE

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): 200MBq of 64Cu-MeCOSar-Octreotate ("64Cu-SARTATE") given as a single bolus intravenous injection.
  Interventions: Drug: 64Cu-SARTATE

INTERVENTIONS:
Drug: 64Cu-SARTATE — 200MBq of 64Cu-MeCOSar-Octreotate ("64Cu-SARTATE") given as a single bolus intravenous injection and peptide mass will not exceed 10micrograms.
  Other Names: 64Cu-MeCOSar-Octreotate

SUMMARY:
The primary purpose of this study is to examine the safety and potential effectiveness of a drug molecule called 64Cu-SARTATE as a potential new way to detect neuroendocrine cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Age greater than or equal to 18 years
3. Life expectancy greater than or equal to 8 weeks
4. Low and Intermediate Grade (Ki-67 index <20%) neuroendocrine tumors (NET)
5. At least one site of active somatostatin receptor positive malignancy, as demonstrated on the pre-study 68Ga-DOTATATE PET/CT scan performed as part of routine clinical care
6. Subjects with an estimated glomerular filtration rate (eGFR) greater than 60ml/min as measured using the MDRD formula (Modification of Diet in Renal Disease).
7. Eastern Cooperative Oncology Group (ECOG) performance score of 0-2

Exclusion Criteria:

1. Pregnant or breastfeeding females
2. Known sensitivity or allergy to somatostatin analogues
3. Subjects who have received interventional treatment for their NET in the interval between 68Ga-DOTATATE PET/CT & 64Cu-SARTATE PET/CT scan
4. Treatment with long acting somatostatin analogues within 28 days prior to the administration of Investigational Product
5. Treatment with short acting somatostatin analogues within 24hrs prior to the administration of Investigational Product
6. QTc interval greater than 0.44seconds as measured by screening ECG
7. Any serious medical condition which the investigator feels may interfere with the procedures or evaluations of the study
8. Patients unwilling or unable to comply with protocol or with a history of non-compliance or inability to grant informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05-21 (Actual); Primary Completion 2016-02-25 (Actual); Study Completion 2016-02-25 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events related to 64Cu-SARTATE | 1 week post administration
  Occurrence of adverse clinical, biochemical or haematological events assessed for up to 1 week post administration of 64Cu-SARTATE.
Percentage of injected 64Cu-SARTATE dose found in organs of interest | At 30 minutes following administration
  Percentage of injected 64Cu-SARTATE dose found in organs of interest via whole body PET scan
Percentage of injected 64Cu-SARTATE dose found in organs of interest | At 1 hour following administration
  Percentage of injected 64Cu-SARTATE dose found in organs of interest via whole body PET scan
Percentage of injected 64Cu-SARTATE dose found in organs of interest | At 4 hours following administration
  Percentage of injected 64Cu-SARTATE dose found in organs of interest via whole body PET scan
Percentage of injected 64Cu-SARTATE dose found in organs of interest | At 24 hours following administration
  Percentage of injected 64Cu-SARTATE dose found in organs of interest via whole body PET scan
Absorbed organ dose | At 30 minutes following administration
  Absorbed organ doses expressed as micro Sv/MBq of administered 64Cu-SARTATE, and whole body dose expressed as milliSv/200MBq of administered dose as assessed using whole body PET scan (composite outcome)
Absorbed organ dose | At 1 hour following administration
  Absorbed organ doses expressed as micro Sv/MBq of administered 64Cu-SARTATE, and whole body dose expressed as milliSv/200MBq of administered dose as assessed using whole body PET scan (composite outcome)
Absorbed organ dose | At 4 hours following administration
  Absorbed organ doses expressed as micro Sv/MBq of administered 64Cu-SARTATE, and whole body dose expressed as milliSv/200MBq of administered dose as assessed using whole body PET scan (composite outcome)
Absorbed organ dose | At 24 hours following administration
  Absorbed organ doses expressed as micro Sv/MBq of administered 64Cu-SARTATE, and whole body dose expressed as milliSv/200MBq of administered dose as assessed using whole body PET scan (composite outcome)

SECONDARY OUTCOMES:
Demonstration of known malignancy | 30 minutes, 1 hour, 4 hours and 24 hours following administration
  Whether 64Cu-SARTATE PET/CT scans demonstrate known sites of 68Ga-DOTATATE avid malignancy with equivalent or greater tumor to background ratios, where background uptake is that found in a non-tumor containing area of interest as decided upon by the nuclear medicine physician at the time of scan assessment.
Uptake in non-physiological, non-tumor containing tissues | 30 minutes, 1 hour, 4 hours and 24 hours following administration
  Whether 64Cu-SARTATE PET/CT scans demonstrate any non-physiological, non-tumor containing tissues with uptake greater than 1.5 x that of the background, where background uptake is defined as in secondary endpoint.

IPD SHARING:
Plan to Share IPD: No